CLINICAL TRIAL: NCT00661609
Title: A Phase II, Single Arm, Single Agent, Multicentre, Adaptive 2-Stage Study to Evaluate the Efficacy, Safety, and Pharmacokinetics of AZD4877 Administered Weekly in Patients With Recurrent Advanced Urothelial Cancer
Brief Title: A Phase II Study of AZD4877 (a Novel Anti-mitotic Agent) in Advanced Bladder Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Jeffrey Skolnik, MD/Associate Medical Director, AstraZeneca
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D2782C00010
Record Dates: First submitted 2008-04-16; First posted 2008-04-18 (Estimated); Results first posted 2011-01-12 (Estimated); Last update posted 2011-01-12 (Estimated); Status verified 2010-12

CONDITIONS: Bladder Cancer; Transitional Cell Bladder Cancer; Urethra Cancer; Ureter Cancer; Renal Pelvis Cancer
Keywords: Anti-mitotic; Eg5 Inhibitor; Kinesin Spindle Protein Inhibitor; Urothelial Cancer; Bladder Cancer; Renal Pelvis Cancer; Urethra Cancer; Ureter Cancer; Recurrent; Advanced; Stage IV
MeSH Terms: conditions — Urinary Bladder Neoplasms; Urethral Neoplasms; Ureteral Neoplasms; Recurrence | interventions — N-(3-aminopropyl)-N-(1-(5-benzyl-3-methyl-4-oxo-(1,2)thiazolo(5,4-d)pyrimidin-6-yl)-2-methylpropyl)-4-methylbenzamide

ARMS (1):
- AZD4877 (Experimental): Single agent AZD4877
  Interventions: Drug: AZD4877

INTERVENTIONS:
Drug: AZD4877 — Intravenous (IV)25mg/weekly

SUMMARY:
The purpose of this Phase II study is to determine if AZD4877, an experimental drug that is a novel anti-mitotic agent (Eg5 or Kinesin Spindle Protein inhibitor that interferes with tumor cell division leading to tumor growth), can reduce tumor sizes in patients with bladder cancer

ELIGIBILITY:
Inclusion Criteria:

* Confirmed urothelial cancer (cancer of the bladder, renal pelvis, ureter, or urethra).
* Tumor, Node, Metastasis (TNM) Stage IV urothelial cancer that can not be helped by curative surgery and/or curative radiotherapy
* Must have had a maximum of 2 prior chemotherapeutic regimens, one for unremovable and/or metastasized disease, and the other in the adjuvant or neo-adjuvant setting.
* Ambulatory and capable of all selfcare more than 50% of waking hours

Exclusion Criteria:

* Prior treatment with investigational or standard anti-cancer agents, including radiotherapy, within 4 weeks prior to first dose of study medication; 6 weeks if prior systemic mitomycin, nitrosourea, or suramin.
* Inadequate bone marrow reserve
* Inadequate liver function in the presence of liver metastases
* Impaired renal function

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2008-05; Primary Completion 2009-05 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gary Hudes, MD, Principal Investigator — Fox Chase Cancer Center
Locations (36):
- United States (18):
  - Research Site, Palo Alto, California
  - Research Site, San Bernardino, California
  - Research Site, Southington, Connecticut
  - Research Site, Miami, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Marietta, Georgia
  - Research Site, Chicago, Illinois
  - Research Site, Scarborough, Maine
  - Research Site, Ann Arbor, Michigan
  - Research Site, Minneapolis, Minnesota
  - Research Site, Hackensack, New Jersey
  - Research Site, Morristown, New Jersey
  - Research Site, New York, New York
  - Research Site, Charlotte, North Carolina
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Woonsocket, Rhode Island
  - Research Site, Seattle, Washington
  - Research Site, Morgantown, West Virginia
- Canada (5):
  - Research Site, Vancouver, British Columbia
  - Research Site, Halifax, Nova Scotia
  - Research Site, Toronto, Ontario
  - Research Site, Montreal, Quebec
  - Research Site, Québec, Quebec
- Germany (5):
  - Research Site, Berlin
  - Research Site, Dresden
  - Research Site, Düsseldorf
  - Research Site, München
  - Research Site, Münster
- Spain (2):
  - Research Site, Barcelona
  - Research Site, Madrid
- United Kingdom (6):
  - Research Site, Leeds, West Yorkshire
  - Research Site, Glasgow
  - Research Site, London
  - Research Site, Manchester
  - Research Site, Southampton
  - Research Site, Surrey

REFERENCES:
- [Derived] Jones R, Vuky J, Elliott T, Mead G, Arranz JA, Chester J, Chowdhury S, Dudek AZ, Muller-Mattheis V, Grimm MO, Gschwend JE, Wulfing C, Albers P, Li J, Osmukhina A, Skolnik J, Hudes G. Phase II study to assess the efficacy, safety and tolerability of the mitotic spindle kinesin inhibitor AZD4877 in patients with recurrent advanced urothelial cancer. Invest New Drugs. 2013 Aug;31(4):1001-7. doi: 10.1007/s10637-013-9926-y. Epub 2013 Jan 18. PMID 23329066

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited at 23 study sites in 5 countries: United States (7 centers), United Kingdom (6 centers), Germany (5 centers), Canada (3 centers), and Spain (2 centers) between 29 May 2008 and 11 January 2010. 54 participants were enrolled into the study of which 41 participants received at least one dose of study medication.
Pre-assignment Details: Following enrolment there was a screening period of up to 28 days, after which if all inclusion/exclusion criteria were met, patients were dosed with AZD4877.
Groups:
- AZD4877: AZD4877 25 mg (Intravenous (IV), 25mg weekly)
Period: Overall Study
Arm/Group | AZD4877
Started | 41 (All dosed patients)
Completed | 0 (Treatment is not for a fixed period and continues until a discontinuation criterion is met.)
Not Completed | 41
Not completed — Adverse Event | 4
Not completed — Death | 20
Not completed — Withdrawal by Subject | 2
Not completed — PI Decision | 1
Not completed — Survival follow up stage discontinued | 11
Not completed — Disease progression | 3

BASELINE CHARACTERISTICS:
Arm/Group | AZD4877
Number analyzed (Participants) | 41
Age, Customized [Number; unit: Participants]
  >=18 - <65 Years | 17
  >=65 - <75 Years | 19
  >=75 Years | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 30
Race/Ethnicity, Customized [Number; unit: participants]
  White | 40
  Black and African | 1

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR) as Evaluated by Response Evaluation Criteria In Solid Tumors (RECIST)
Description: Percentage of participants with complete response (CR) or partial response (PR) as per Response Evaluation Criteria In Solid Tumors (RECIST), version 1.0 (Therasse et al. Natl Cancer Inst 92 (2000) pp205-216).
Time Frame: 8 weeks after study drug begins & and every 8 wks thereafter until discontinuation of study drug ( maximum treatment period of 309 days (44 weeks)
Population: Of the 41 participants who received at least one dose of study medication, only 39 were evaluable for response by RECIST (excludes 2 patients who had baseline scans performed more than 28 days before dosing).
Measure: Number; unit: Percengate of participants
Arm/Group | AZD4877
Number analyzed (Participants) | 39
Percengate of participants | 2.6

2. Secondary Outcome: Disease Control Rate (DCR)
Description: Percentage of participants with Complete Response (CR), Partial Response (PR), or stable disease (SD) lasting at least 8 weeks from the first administration of study drug. RECIST guidelines:(Response evaluation criteria in solid tumors, version 1.0).
Time Frame: 8 weeks after study drug begins & every 8 weeks thereafter until discontinuation of the study ( maximum treatment period of 309 days (44 weeks)
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | AZD4877
Number analyzed (Participants) | 39
Percentage of participants | 20.5

3. Secondary Outcome: Duration of Objective Tumor Response (OTR)
Description: Time in weeks from the date of Complete Response (CR) or Partial Response (PR), whichever occurs earlier, to the date of discontinuation of study. RECIST guidelines:(Response evaluation criteria in solid tumors, version 1.0)
Time Frame: Time from first documentation of Complete or Partial Response, whichever occurs earlier, to discontinuation of the study drug (maximum treatment period of 309 days (44 weeks)
Reporting Status: Not Posted
Measure: Number; unit: Time in weeks

4. Secondary Outcome: Progression Free Survival (PFS)
Description: Time in weeks from date of first study drug administration to the date of progressive disease according to the RECIST guidelines (Response evaluation in solid tumors, version 1.0), or death due to any cause.
Time Frame: Time from the first administration of study drug to disease progression or death (maximum treatment period of 309 days (44 weeks)
Population: as for outcome 1
Measure: Median (Full Range); unit: Weeks
Arm/Group | AZD4877
Number analyzed (Participants) | 39
Weeks | 7.3 [0 to 44]

5. Secondary Outcome: Overall Survival (OS)
Description: Time in weeks from the first administration of study drug to death.
Time Frame: as for outcome 4
Population: as for outcome 1
Measure: Median (Full Range); unit: Weeks
Arm/Group | AZD4877
Number analyzed (Participants) | 39
Weeks | 23.1 [1.3 to 48.1]

ADVERSE EVENTS:
Arm/Group | AZD4877
Serious Adverse Events (participants affected / at risk) | 14/41
Other Adverse Events (participants affected / at risk) | 38/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AZD4877 (N=41)
Leukopenia (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 1
Acute Myocardial Infarction (Cardiac disorders) | 1
Cardiac Failure Congestive (Cardiac disorders) | 1
Ventricular Arrhythmia (Cardiac disorders) | 1
Abdominal Pain (Gastrointestinal disorders) | 1
Chest Pain (General disorders) | 1
Death (General disorders) | 1
Fatigue (General disorders) | 1
Urinary Tract Infection (Infections and infestations) | 2
Infection (Infections and infestations) | 1
Narcotic Intoxication (Injury, poisoning and procedural complications) | 1
Dehydration (Metabolism and nutrition disorders) | 2
Mental Status Changes (Psychiatric disorders) | 1
Haematuria (Renal and urinary disorders) | 1
Renal Failure Acute (Renal and urinary disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AZD4877 (N=41)
Neutropenia (Blood and lymphatic system disorders) | 23
Anaemia (Blood and lymphatic system disorders) | 11
Leukopenia (Blood and lymphatic system disorders) | 7
Nausea (Gastrointestinal disorders) | 11
Constipation (Gastrointestinal disorders) | 8
Vomiting (Gastrointestinal disorders) | 8
Abdominal Pain (Gastrointestinal disorders) | 5
Diarrhoea (Gastrointestinal disorders) | 5
Abdominal Discomfort (Gastrointestinal disorders) | 3
Abdominal Distension (Gastrointestinal disorders) | 3
Fatigue (General disorders) | 13
Pyrexia (General disorders) | 7
Asthenia (General disorders) | 5
Influenza Like Illness (General disorders) | 4
Oedema Peripheral (General disorders) | 4
Urinary Tract Infection (Infections and infestations) | 11
Oral Candidiasis (Infections and infestations) | 3
Weight Decreased (Infections and infestations) | 5
Anorexia (Metabolism and nutrition disorders) | 7
Back Pain (Musculoskeletal and connective tissue disorders) | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 3
Groin Pain (Musculoskeletal and connective tissue disorders) | 3
Neck Pain (Musculoskeletal and connective tissue disorders) | 3
Headache (Nervous system disorders) | 4
Lethargy (Nervous system disorders) | 4
Insomnia (Psychiatric disorders) | 5
Haematuria (Renal and urinary disorders) | 3
Pollakiuria (Renal and urinary disorders) | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
An Investigator agrees to provide a copy of the publication to AZ for review at least 60 days in advance of submission for publication. Investigators in multicenter (MC) studies agree to postpone MC publications until the earlier of the date of the first AZ-authorized MC publication or a period up to 18 months from study completion at all sites. AZ has the right to request delays: up to 60 days for confidential information, and an additional 90 days to protect intellectual property.